CLINICAL TRIAL: NCT04864158
Title: Prosthesis Versus Active Exercise Program in Patients With Rotator Cuff Arthropathy Eligible For Reverse Shoulder Arthroplasty: the ReAct Multicenter, Randomized Controlled Trial
Brief Title: Prosthesis Versus Active Exercise Program in Patients With Rotator Cuff Arthropathy
Acronym: REACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Tampere University Hospital (Other); Aalborg University Hospital (Other); Regionshospitalet Silkeborg (Other); Oslo University Hospital (Other); The Danish Rheumatism Association (Other); Association of Danish Physiotherapists (Other); Regionshospitalet Viborg, Skive (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Tartu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REACT
Record Dates: First submitted 2021-04-13; First posted 2021-04-28 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff Arthropathy
Keywords: Physiotherapist-supervised Exercise; Physical Therapy; Physical Rehabilitation; Reverse Shoulder Arthroplasty; Randomized Controlled Trial; Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSA-group (Experimental): Surgery
  Interventions: Procedure: TSA-group
- Exercise-group (Experimental): Exercise
  Interventions: Other: Exercise-group

INTERVENTIONS:
Procedure: TSA-group — Reverse total shoulder arthroplasty followed by standard rehabilitation.
  Arms: RSA-group
Other: Exercise-group — The exercise-group will attend a 12-week exercise program with one weekly physiotherapist-supervised session supplemented with two weekly sessions of home-based exercises. Utilisation of a predefined training protocol describing procedures and content of each session secure uniformity and standardisation of the intervention. The exercise program consists of two warm-up exercises and five exercises that target shoulder range of motion and muscle strength. Furthermore, a link to a video, informing about glenohumeral osteoarthritis, the role of exercise and exercise related pain, will be sent to all patients in the exercise-group. The physiotherapists delivering the exercise intervention are not otherwise related to the trial.
  Arms: Exercise-group

SUMMARY:
Reverse shoulder arthroplasty (RSA) is a well-established treatment for rotator cuff arthropathy. However, the effectiveness of RSA has not been compared to non-surgical treatment in a randomised controlled trial. Shoulder exercises may be an effective treatment for reducing pain and improving function in glenohumeral osteoarthritis. The primary aim of this trial is to examine if RSA followed by standard postsurgical rehabilitation is superior to a 12-week exercise programme in patients with rotator cuff arthropathy eligible for unilateral RSA. The investigators hypothesise that surgical intervention followed by standard rehabilitation, results in clinically relevant (14-point, on a scale from 0-100) improvement compared to the exercise intervention.

DETAILED DESCRIPTION:
Rotator cuff arthropathy describes the clinical scenario of massive rotator cuff ruptures associated with glenohumeral joint degeneration and superior migration of the humeral head. Clinical presentation includes joint effusion, pain, and loss of mobility. Reverse shoulder arthroplasty (RSA) is a well-established treatment for rotator cuff arthropathy. Several studies have suggested the need for trials comparing shoulder arthroplasty to non-surgical treatments.

The ProAct trial is a Nordic multicenter randomized controlled trial. Patients with rotator cuff arthropathy, eligible for a RSA will be randomised to either RSA followed by usual care or exercise only. The exercise intervention consists of 12 weeks of exercise with one weekly physiotherapist-supervised exercise session.

The primary outcome will be the total the Western Ontario Osteoarthritis of the Shoulder index score at 12 months follow-up. Outcome assessment will be performed at baseline, and at 3 and 12 months and 2-, 5- and 10 years after start of surgical/non-surgical treatment.

Patients fulfilling the eligibility criteria but declining to participate in the randomised trial will be offered the option of participating in an observational cohort using the same primary end point and patient reported outcomes, but following usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60-85 years
* Eligible for RSA
* Rotator cuff arthropathy according to Hamada grade 3, 4 and 5 (33)

Exclusion Criteria:

* Previous shoulder fracture (fracture of the proximal humerus or glenoid fracture)
* Planned other upper extremity surgery within six months
* Rheumatoid arthritis or other types of arthritis not diagnosed as primary glenohumeral OA
* Cancer diagnosis and receiving chemo-, immuno- or radiotherapy
* Neurological diseases affecting shoulder mobility (e.g. disability after previous stroke, multiple sclerosis, Parkinson's, Alzheimer's disease)
* Other reasons for exclusion (i.e. mentally unable to participate) or planned absence for more than 14 days in the first 3 months after baseline test.
* Unable to communicate in the participating countries respective languages

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2038-11 (Estimated)

PRIMARY OUTCOMES:
the Western Ontario Osteoarthritis of the Shoulder index (WOOS) | Measured at 12 month follow-up
  WOOS consist of 19 items to be answered using a visual analog scale (VAS). Each item has a possible score ranging from 0 to 100, leading to a total WOOS score ranging from 0 to 1900, with 0 being the best. For simplicity reasons, raw scores can be converted to a percentage of the maximum score (0-100, 100 best).

SECONDARY OUTCOMES:
the Western Ontario Osteoarthritis of the Shoulder index (WOOS) | Measured at baseline, 12-week, 2-, 5- and 10-year follow-up
  WOOS consist of 19 items to be answered using a visual analog scale (VAS). Each item has a possible score ranging from 0 to 100, leading to a total WOOS score ranging from 0 to 1900, with 0 being the best. For simplicity reasons, raw scores can be converted to a percentage of the maximum score (0-100, 100 best).
Disabilities of the Arm, Shoulder and Hand (DASH) | Measured at baseline, 12-week, 12-month, 2-, 5- and 10-year follow-up
  DASH is a self-administered questionnaire that consist of thirty core items and eight items assessing work and sports and/or performing arts activities. Each individual item is scored on a 5-point Likert scale, and lower scores correlated to minimal impairments and higher scores indicate more impairment. The cumulative DASH score is scaled from 0-100 with higher scores indicating more disability
The change in pain measured on a 100 mm Visual Analogue Scale (VAS) | Measured at baseline, 12-week, 12-month, 2-, 5- and 10-year follow-up
  Patient reported pain intensity at rest, during activity and nightly pain. With a possible score ranging from 0 to 100, with 100 indicating the worst possible pain
The use of analgesics during the last week | Measured at baseline, 12-week, 12-month, 2-, 5- and 10-year follow-up
  The patients will be asked if they take any analgesics (yes/no)
The type of analgesics consumed during the last week | Measured at baseline, 12-week, 12-month, 2-, 5- and 10-year follow-up
  The patients will be asked which type of analgesics they take (paracetamol, NSAID, morphine/opioids).
Consumption of analgesics during the last week | Measured at baseline, 12-week, 12-month, 2-, 5- and 10-year follow-up
  The patients will be asked how often they consume the analgesic medication (never, daily, weekly, monthly).
Serious Adverse Events | The patients in the surgical intervention group will be monitored for serious adverse events during the 4 weeks from the discharge.
  Serious adverse events are defined as embolism (cardiac or brain), death, liver and renal failure.
Adverse events | Occurring during the period from inclusion until the 12-month follow-up
  Defined as any unintended and unfavorable sign, symptom or disease resulting in contact with the healthcare system irrespective of a causal relationship with the intervention and outcome assessments.

OTHER OUTCOMES:
Accelerometer-based activity using tri-axial (Axivity, UK) accelerometers | Measured at baseline and 12-month follow-up
  The patients will have an accelerometer sensor mounted with tape to both upper arms for 4 days. The sensors will measure 24/7 activity of the upper arms.
Accelerometer-based degree of movement using tri-axial (Axivity, UK) accelerometers | Measured at baseline and 12-month follow-up
  The patients will have an accelerometer sensor mounted with tape to both upper arms for 4 days. The sensors will measure 24/7 degree of movement.
The 100 mm Visual Analogue Scale (exercise-group) | Measured immediately before and immideately after each exercise session. From the date of the start of the exercise intervention until the end of the exercise intervention, assessed up to 12 months.
  Patient reported pain intensity at rest. With a possible score ranging from 0 to 100, with 100 indicating the worst possible pain.
EuroQol Group 5-dimension 5-level (EQ-5D-5L) | Measured at baseline, 12-week, 12-month, 2- 5- and 10-year follow-up.
  The EuroQol measures the five dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each dimension consists of one item, distinguished in five levels. We will used the UK value set in this study, because a Danish value set is not yet available. These values range from -0.285 to 1.0, a value of 1.0 corresponds to full health, 0 corresponds to death and negative values correspond to health status considered to be worse than death.
Productivity Costs Questionnaire (iPCQ) | Measured at 12-week and 12-month.
  The iPCQ is a questionnaire for the measurement of costs in economic evaluations. It consists of 18 questions of which 9 are general questions followed by questions to measure productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work. The minimum value is 0 (no productivity loss) and the maximum value is infinite. Measured for the health economic evaluation in Denmark.
Patient Acceptable Symptom State (PASS) | Measured at 12-month, 2-, 5- and 10-year follow-up.
  PASS will be assessed with the following question, reported by the patient: "When you think of your shoulder function, will you consider your current condition as satisfying? By shoulder function, you should take into account your activities of daily living, sport and recreational activities, your shoulder pain and other symptoms and your quality-of-life", measured on a dichotomous scale (yes/no).
Treatment Failure | Measured at 12-month, 2-, 5- and 10-year follow-up.
  Patient-reported treatment failure will be assessed only by patients answering "no" to PASS with the following question: "Would you consider your current state as being so unsatisfactory that you think the treatment has failed?" on a dichotomous scale (yes/no).
Number of total shoulder arthroplasty surgeries (exercise-group) | Measured from baseline to 12-month, 2-, 5- and 10-year follow-up.
  Number of total shoulder arthroplasty surgeries performed in the exercise-group.
Number of supervised exercise sessions from baseline to 3 months (exercise-group) | From baseline to 12-week
  High compliance will be defined as participation in ≥70 percent of the training sessions; moderate compliance as participation in 50-70 percent of the sessions; and poor compliance as participation in <50 percent of the sessions.
Number of patients performing unsupervised exercise (exercise-group) | From baseline to 12-week
  Adherence to two weekly unsupervised exercise sessions will be measured by a patient-reported questionnaire
Number of patients performing unsupervised exercise (exercise-group) | From 12-week to 12-month
  Adherence to optional unsupervised exercise sessions will be measured by a patient-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Josefine B. Larsen, MSc, Principal Investigator — Aarhus University Hospital and Aarhus University; Inger Mechlenburg, Prof., Study Director — Aarhus University Hospital and Aarhus University; Theis M. Thillemann, PhD, As Prof, Study Director — Aarhus University Hospital and Aarhus University; Antti P. Launonen, PhD, As Prof, Study Director — Tampere University Hospital
Locations (8):
- Denmark (5):
  - Aarhus University Hospital, Aarhus N
  - Esbjerg Hospital, Esbjerg
  - Aalborg University Hospital, Farsø
  - Silkeborg Regional Hospital, Silkeborg
  - Viborg Regional Hospital, Viborg
- Tartu University Hospital, Tartu, Estonia
- Tampere University Hospital, Tampere, Finland
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Pseudo anonymised patient-level data for the primary and all secondary outcome measures will be made available if required by the scientific journal, in which the results of the trial are published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial
Access Criteria: Data access will be reviewed by the author group. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Larsen JB, Thillemann TM, Launonen AP, Ostergaard HK, Falstie-Jensen T, Reito A, Jensen SL, Mechlenburg I. Prosthesis versus exercise for rotator cuff tear arthropathy - protocol of a randomised controlled trial. Dan Med J. 2025 Aug 22;72(9):A09240645. doi: 10.61409/A09240645. PMID 40927835